CLINICAL TRIAL: NCT00001016
Title: A Treatment Protocol for the Use of Trimetrexate With Leucovorin Rescue for AIDS Patients With Pneumocystis Carinii Pneumonia and Serious Intolerance to Approved Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: TX 301
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 1993-07

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimetrexate; Pneumonia, Pneumocystis carinii; Quinazolines; Infusions, Intravenous; Injections, Intravenous; Leucovorin; Drug Evaluation; Drug Therapy, Combination; Administration, Oral; Acquired Immunodeficiency Syndrome; Antiprotozoal Agents; AIDS-Related Complex
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — trimetrexate glucuronate; Leucovorin

INTERVENTIONS:
Drug: Trimetrexate glucuronate
Drug: Leucovorin calcium

SUMMARY:
To determine the safety and effectiveness of an investigational drug trimetrexate (TMTX) with leucovorin rescue (LCV) in the treatment of Pneumocystis carinii pneumonia (PCP) in patients who have AIDS, are HIV positive, or are at high risk for HIV infection, and who have demonstrated serious adverse effects from the conventional therapies for PCP.

The drugs usually used to treat PCP in AIDS patients (trimethoprim / sulfamethoxazole and pentamidine) have had to be discontinued in many patients because of severe adverse effects. Currently there are no proven alternatives to these drugs. TMTX was chosen for this trial because it has been found to be very active against the PCP organism in laboratory tests. In a preliminary trial, TMTX in combination with LCV has been effective against PCP with fewer and less severe adverse effects.

DETAILED DESCRIPTION:
The drugs usually used to treat PCP in AIDS patients (trimethoprim / sulfamethoxazole and pentamidine) have had to be discontinued in many patients because of severe adverse effects. Currently there are no proven alternatives to these drugs. TMTX was chosen for this trial because it has been found to be very active against the PCP organism in laboratory tests. In a preliminary trial, TMTX in combination with LCV has been effective against PCP with fewer and less severe adverse effects.

AMENDED: 08/01/90. As of August 31, 1989, 437 patients were enrolled into uncontrolled studies of trimetrexate for PCP:214 in TX 301/ACTG 0=039 (trimetrexate for patients intolerant of approved therapies) and 223 in NS 401 (trimetrexate for patients refractory to approved therapies). The analysis of overall response rate, stringently defined as having received at least 14 days of trimetrexate and being alive at follow-up 1 month after the completion of therapy, reveals 84/159 intolerant patients and 48/160 refractory patients had responded, for rates of 53 percent and 30 percent, respectively. These response rates include all individuals who received at least one dose of trimetrexate. Of the 111 patients who were ventilator-dependent at study entry, 18 completed a course of therapy and were alive a month later, for a response rate of 16 percent. All other ventilated patients died. The most common severe (grades 3 and 4) toxicities were: transaminase elevation (greater than 5 x normal) in 94 patients, anemia (less than 7.9 g/dl) in 109, neutropenia (less than 750 cells/mm3) in 58, fever (greater than 40 degrees C) in 37, and thrombocytopenia (less than 50,000 platelets/mm3) in 27.

Toxicity required discontinuation of therapy in approximately 5 percent of all patients. Original design: Patients entered in the study are given TMTX once a day for 21 days and LCV 4 times a day (every 6 hours) for 24 days. Doses are determined by body size. Both drugs are given by intravenous infusion, but LCV may be given orally after the first 10 days. Doses are adjusted if side effects, such as low white blood cell counts, are too severe. During the 21-day trial, zidovudine (AZT) may not be used because of possible increased bone marrow toxicity. AZT may be resumed as soon as the administration of TMTX and LCV has been completed. After treatment with TMTX, the patient may be treated with other drugs to prevent the recurrence of PCP at the discretion of his/her physician.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Blood pressure medication.

Concurrent Treatment:

Allowed:

* Blood products.
* Ventilatory support.

Patients must have the following:

* Diagnosis of Pneumocystis carinii pneumonia (PCP).
* Be HIV positive by ELISA, HIV culture, or p24 antigenemia; or be a member of an identified risk group.
* Intolerant to trimethoprim / sulfamethoxazole (TMP / SMX).
* Intolerant to pentamidine.

Prior Medication:

Allowed:

* Trimethoprim / sulfamethoxazole trials.
* Pentamidine trials.
* Myelosuppressive agents.
* Nephrotoxic agents.
* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients who do not meet the inclusion criteria are excluded.

Concurrent Medication:

Excluded:

* Myelosuppressive agents.
* Nephrotoxic agents.
* Other investigational drugs including high-dose steroids (exceeding physiologic replacement doses).

Patients who do not meet the inclusion criteria are excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feinberg J, Study Chair
Locations (1):
- Warner-Lambert Parke-Davis, Morris Plains, New Jersey, United States